CLINICAL TRIAL: NCT02596035
Title: A Phase 3b/4 Safety Trial of Nivolumab (BMS-936558) in Subjects With Advanced or Metastatic Renal Cell Carcinoma (CheckMate 374: CHECKpoint Pathway and Nivolumab Clinical Trial Evaluation 374)
Brief Title: An Investigational Immuno-therapy Safety Trial of Nivolumab in Patients With Advanced or Metastatic Renal Cell Carcinoma
Acronym: CheckMate 374
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CA209-374; 2015-003286-28 (EudraCT Number)
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab dose as specified
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab
  Other Names: Opdivo

SUMMARY:
This study will generate safety data on Nivolumab given by itself in treatment of advanced Renal Cell Carcinoma (RCC). The primary objective of this study is to assess immune related side effects, also known as immune-mediated adverse events (IMAEs), in patients treated with Nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or Metastatic renal cell carcinoma (RCC)
* Predominant clear cell histology:

  1. At least 1 but no more than 2 prior systemic anti vascular endothelial growth factor (anti-VEGF) treatments
  2. No more than 3 total prior systemic treatment regimens in the advanced or metastatic setting
  3. Subjects with prior treatment with a mechanistic target of rapamycin (mTOR) are eligible
* Non-clear cell histology: 0-3 prior systemic therapies and may include mTOR inhibitor
* Brain metastases allowed if asymptomatic, without edema, and not receiving corticosteroids or radiation
* Performance Status (PS): ≥ 70% Karnofsky Performance Scale (KPS)
* All Memorial Sloan-Kettering Cancer Center (MSKCC) prognostic scores allowed

Exclusion Criteria:

* Subjects with any active autoimmune disease or a history of known autoimmune disease
* History of severe hypersensitivity reaction to other monoclonal antibodies
* Prior malignancy, active within the last 3 years, except for locally curable cancers which have been apparently cured
* Known HIV or AIDS-related illness
* Any positive tests for Hepatitis B or Hepatitis C virus indicating acute or chronic infection

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (39):
- United States (39):
  - Local Institution - 0030, Phoenix, Arizona
  - Comprehensive Blood And Cancer Center, Bakersfield, California
  - St. Jude Hospital Yorba Linda, Fullerton, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Sansum Santa Barbara Medical Foundation Clinic, Santa Barbara, California
  - University Of Colorado, Aurora, Colorado
  - Local Institution - 0028, Grand Junction, Colorado
  - Local Institution - 0018, Lakewood, Colorado
  - Local Institution - 0008, Fort Myers, Florida
  - Baptist Health Medical Group Oncology, Miami, Florida
  - Local Institution - 0007, St. Petersburg, Florida
  - Local Institution - 0054, Tampa, Florida
  - Illinois Cancer Specialists, Niles, Illinois
  - Local Institution - 0052, Fort Wayne, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - HCA Midwest Division, Kansas City, Missouri
  - Southeast Nebraska Hematology & Oncology Consultants, P.C., Lincoln, Nebraska
  - Local Institution - 0011, Omaha, Nebraska
  - Urology Cancer Center Laboratory, Omaha, Nebraska
  - Local Institution - 0014, Las Vegas, Nevada
  - Local Institution - 0053, Buffalo, New York
  - Broome Oncology, Johnson City, New York
  - Local Institution - 0055, New York, New York
  - Local Institution - 0001, Tulsa, Oklahoma
  - Local Institution - 0016, Portland, Oregon
  - Local Institution - 0020, Charleston, South Carolina
  - Local Institution - 0005, Chattanooga, Tennessee
  - Local Institution - 0012, Germantown, Tennessee
  - Local Institution - 0004, Nashville, Tennessee
  - Local Institution - 0015, Dallas, Texas
  - The Center For Cancer And Blood Disorders, Fort Worth, Texas
  - Local Institution - 0034, Houston, Texas
  - Local Institution - 0021, San Antonio, Texas
  - Texas Cancer Center - Sherman, Sherman, Texas
  - Local Institution - 0032, Norfolk, Virginia
  - Local Institution - 0047, Richmond, Virginia
  - Local Institution - 0017, Roanoke, Virginia
  - Local Institution - 0039, Seattle, Washington

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 142 Participants were treated
Groups:
- Clear Cell Histology: Participants with predominant clear cell histology received Nivolumab at a dose of 240 mg Q2W by a 30-minute IV infusion.
- Non-Clear Cell Histology: Participants with non-clear cell histology received Nivolumab at a dose of 240 mg Q2W by a 30-minute IV infusion.
- Brain Metastasis: Participants with brain metastases regardless of histology received Nivolumab at a dose of 240 mg Q2W by a 30-minute IV infusion.
Period: Overall Study
Arm/Group | Clear Cell Histology | Non-Clear Cell Histology | Brain Metastasis
Started | 97 | 44 | 1
Completed | 0 | 0 | 0
Not Completed | 97 | 44 | 1
Not completed — Disease Progression | 64 | 32 | 1
Not completed — study drug toxicity | 12 | 3 | 0
Not completed — AE unrelated to study drug | 5 | 2 | 0
Not completed — participant request to discontinue study treatment | 2 | 0 | 0
Not completed — participant withdrew consent | 2 | 2 | 0
Not completed — Poor/Non Comlpiance | 0 | 1 | 0
Not completed — participant no longer meets study criteria | 1 | 0 | 0
Not completed — other reasons | 11 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clear Cell Histology | Non-Clear Cell Histology | Brain Metastasis | Total
Number analyzed (Participants) | 97 | 44 | 1 | 142
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (10.33) | 61.4 (12.88) | 32 (NA) — Only 1 participant was evaluable in this arm. | 63.5 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 12 | 1 | 44
  Male | 66 | 32 | 0 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 4 | 1 | 16
  Not Hispanic or Latino | 86 | 39 | 0 | 125
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 8 | 0 | 13
  White | 90 | 34 | 1 | 125
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced High-Grade (Grade 3-4 and Grade 5) Immune Mediated Adverse Events (IMAEs)
Description: IMAEs were tabulated using worst grade per Common Terminology Criteria for Adverse Events, National Cancer Institute (NCI CTCAE) Version 4.0 criteria by system organ class and MedDRA version 20.1 preferred term.
Time Frame: Up to 100 days of the last dose of study drug (Approximately 2 years)
Population: Analysis was performed in all treated participants who received any dose of nivolumab.
Measure: Number; unit: Percentage of participants
Arm/Group | Clear Cell Histology | Non-Clear Cell Histology | Brain Metastasis
Number analyzed (Participants) | 97 | 44 | 1
Percentage of participants
  Hepatitis (Grade 3-4) | 4.1 | 0 | 0
  Hepatitis (Grade 5) | 0 | 0 | 0
  Adrenal Insufficiency (Grade 3-4) | 1 | 0 | 0
  Adrenal Insufficiency (Grade 5) | 0 | 0 | 0
  Nephritis And Renal Dysfunction (Grade 3-4) | 1 | 0 | 0
  Nephritis And Renal Dysfunction (Grade 5) | 0 | 0 | 0
  Rash (Grade 3-4) | 1 | 0 | 0
  Rash (Grade 5) | 0 | 0 | 0
  Diabetes mellitus (Grade 3-4) | 3.1 | 0 | 0
  Diabetes mellitus (Grade 5) | 0 | 0 | 0
  Hypothyroidism (Grade 3-4) | 0 | 0 | 0
  Hypothyroidism (Grade 5) | 0 | 0 | 0
  Hypophysitis (Grade 3-4) | 0 | 0 | 0
  Hypophysitis (Grade 5) | 0 | 0 | 0
  Pneumonitis (Grade 3-4) | 0 | 0 | 0
  Pneumonitis (Grade 5) | 0 | 0 | 0
  Hypersensitivity (Grade 3-4) | 0 | 0 | 0
  Hypersensitivity (Grade 5) | 0 | 0 | 0
  Diarrhea/Colitis (Grade 3-4) | 1 | 0 | 0
  Diarrhea/Colitis (Grade 5) | 0 | 0 | 0
  Hyperthyroidism (Grade 3-4) | 0 | 0 | 0
  Hyperthyroidism (Grade 5) | 0 | 0 | 0

2. Secondary Outcome: Median Time to Onset of High Grade (Grade 3-5) Immune Mediated Adverse Events
Description: Time to onset was calculated from first dosing date to the event onset date. If a participant never experienced the given AE, the participant will be censored at the last contact date.
Time Frame: Up to 100 days of the last dose of study drug (Approximately 10 months up to 26 months)
Population: Analysis was performed in all treated participants who received any dose of nivolumab. Here, 'number analyzed' signifies those participants who were evaluable for specified categories.
Measure: Median (Full Range); unit: Days
Arm/Group | Clear Cell Histology | Non-Clear Cell Histology | Brain Metastasis
Number analyzed (Participants) | 97 | 44 | 1
Days
  Adrenal Insufficiency: number analyzed (Participants) | 1 | 0 | 0
  Adrenal Insufficiency | 76.0 [76 to 76] |  |
  Diabetes Mellitus: number analyzed (Participants) | 2 | 0 | 0
  Diabetes Mellitus | 89.0 [46 to 805] |  |
  Hepatitis: number analyzed (Participants) | 4 | 0 | 0
  Hepatitis | 84.5 [47 to 448] |  |
  Nephritis And Renal Dysfunction: number analyzed (Participants) | 1 | 0 | 0
  Nephritis And Renal Dysfunction | 43.0 [43 to 43] |  |
  Rash: number analyzed (Participants) | 1 | 0 | 0
  Rash | 7.0 [7 to 7] |  |
  Diarrhea/Colitis: number analyzed (Participants) | 97 | 0 | 0
  Diarrhea/Colitis | 645.0 [645.0 to 645.0] |  |

3. Secondary Outcome: Median Time to Resolution of High Grade (Grade 3-5) Immune Mediated Adverse Events
Description: Time-to resolution of grade 3-5 AE was defined as the longest time from onset to complete resolution or improvement to the grade at baseline among all clustered select AEs in the category experienced by the participant. Events which worsened into grade 5 events (death) or have a resolution date equal to the date of death are considered unresolved. If a clustered AE is considered as unresolved, the resolution date will be censored to the last known date alive.
Time Frame: From onset of grade 3-5 IMAEs to resolution of IMAEs (Approximately 4 years and 7 months)
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Clear Cell Histology | Non-Clear Cell Histology | Brain Metastasis
Number analyzed (Participants) | 97 | 44 | 1
Days
  Hepatitis: number analyzed (Participants) | 4 | 0 | 0
  Hepatitis | 31.5 [15 to 75] |  |
  Nephritis And Renal Dysfunction: number analyzed (Participants) | 3 | 0 | 0
  Nephritis And Renal Dysfunction | 22.0 [6 to 54] |  |
  Rash: number analyzed (Participants) | 1 | 0 | 0
  Rash | 23.0 [23 to 23] |  |
  Diarrhea/Colitis: number analyzed (Participants) | 1 | 0 | 0
  Diarrhea/Colitis | 154.0 [154 to 154] |  |
  Adrenal Insufficiency: number analyzed (Participants) | 1 | 0 | 0
  Adrenal Insufficiency | NA [NA to NA] — 0 Participants Resolved |  |

4. Secondary Outcome: Percentage of Participants Who Receive Immune Modulating Medication for the Immune-Mediated Event (Any Grade)
Description: Immune modulating medication includes corticosteroids, infliximab, cyclophosphamide, Intravenous immunoglobulin (IVIG), and mycophenolate mofetil
Time Frame: Up to 100 days of the last dose of study drug (Approximately 3 years and 2 months)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Clear Cell Histology | Non-Clear Cell Histology | Brain Metastasis
Number analyzed (Participants) | 97 | 44 | 1
Percentage of participants
  Participants with Pneumonitis: number analyzed (Participants) | 3 | 3 | 0
  Participants with Pneumonitis | 66.7 | 0 |
  Participants with Diarrhea/Colitis: number analyzed (Participants) | 19 | 8 | 0
  Participants with Diarrhea/Colitis | 5.3 | 0 |
  Participants with Hepatitis: number analyzed (Participants) | 12 | 2 | 0
  Participants with Hepatitis | 41.7 | 0 |
  Participants with Adrenal Insufficiency: number analyzed (Participants) | 1 | 0 | 0
  Participants with Adrenal Insufficiency | 100 |  |
  Participants with Nephritis And Renal Dysfunction: number analyzed (Participants) | 22 | 3 | 0
  Participants with Nephritis And Renal Dysfunction | 13.6 | 33.3 |
  Participants with Rash: number analyzed (Participants) | 31 | 8 | 0
  Participants with Rash | 38.7 | 25.0 |
  Participants with Hypersensitivity: number analyzed (Participants) | 3 | 0 | 0
  Participants with Hypersensitivity | 66.7 |  |
  Participants with Hyperthyroidism: number analyzed (Participants) | 8 | 2 | 0
  Participants with Hyperthyroidism | 12.5 | 0 |
  Participants with Hypophysitis: number analyzed (Participants) | 0 | 1 | 0
  Participants with Hypophysitis |  | 100.0 |

5. Secondary Outcome: Percentage of Participants Who Receive More Than Equal to (>=) 40 mg Prednisone Equivalents for the Immune-Mediated Event
Description: as for outcome 4
Time Frame: Up to 100 days of the last dose of study drug (Approximately 3 years and 2 months)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Clear Cell Histology | Non-Clear Cell Histology | Brain Metastasis
Number analyzed (Participants) | 97 | 44 | 1
Percentage of participants
  Participants with Pneumonitis: number analyzed (Participants) | 3 | 3 | 0
  Participants with Pneumonitis | 66.7 | 0 |
  Participants with Diarrhea/Colitis: number analyzed (Participants) | 19 | 8 | 0
  Participants with Diarrhea/Colitis | 5.3 | 0 |
  Participants with Hepatitis: number analyzed (Participants) | 12 | 2 | 0
  Participants with Hepatitis | 41.7 | 0 |
  Participants with Adrenal Insufficiency: number analyzed (Participants) | 1 | 0 | 0
  Participants with Adrenal Insufficiency | 0 |  |
  Participants with Nephritis And Renal Dysfunction: number analyzed (Participants) | 22 | 3 | 0
  Participants with Nephritis And Renal Dysfunction | 9.1 | 0 |
  Participants with Rash: number analyzed (Participants) | 31 | 8 | 0
  Participants with Rash | 6.5 | 0 |
  Participants with Hypersensitivity: number analyzed (Participants) | 3 | 0 | 0
  Participants with Hypersensitivity | 66.7 |  |
  Participants with Hyperthyroidism: number analyzed (Participants) | 8 | 2 | 0
  Participants with Hyperthyroidism | 12.5 | 0 |
  Participants with Hypophysitis: number analyzed (Participants) | 0 | 1 | 0
  Participants with Hypophysitis |  | 100.0 |

6. Secondary Outcome: Total Duration of All Immune Modulating Medications Given for the Immune-Mediated Event
Description: as for outcome 4
Time Frame: From the initiation of Immune modulating medication to discontinuation (approximately 4 years and 9 months).)
Population: as for outcome 2
Measure: Median (Full Range); unit: Weeks
Arm/Group | Clear Cell Histology | Non-Clear Cell Histology | Brain Metastasis
Number analyzed (Participants) | 97 | 44 | 1
Weeks
  Pneumonitis: number analyzed (Participants) | 2 | 0 | 0
  Pneumonitis | 111.07 [8.1 to 214.0] |  |
  Diarrhea/Colitis: number analyzed (Participants) | 1 | 0 | 0
  Diarrhea/Colitis | 7.9 [7.9 to 7.9] |  |
  Hepatitis: number analyzed (Participants) | 5 | 0 | 0
  Hepatitis | 7.00 [1.4 to 230.3] |  |
  Adrenal Insufficiency: number analyzed (Participants) | 1 | 0 | 0
  Adrenal Insufficiency | 241.14 [241.14 to 241.14] |  |
  Nephritis And Renal Dysfunction: number analyzed (Participants) | 3 | 1 | 0
  Nephritis And Renal Dysfunction | 1.14 [0.1 to 7.4] | 1.9 [1.9 to 1.9] |
  Rash: number analyzed (Participants) | 12 | 2 | 0
  Rash | 9.29 [2.1 to 93.9] | 137.43 [17.6 to 257.3] |
  Hypersensitivity: number analyzed (Participants) | 2 | 0 | 0
  Hypersensitivity | 0.1 [0.1 to 0.1] |  |
  Hyperthyroidism: number analyzed (Participants) | 1 | 0 | 0
  Hyperthyroidism | 8.4 [8.4 to 8.4] |  |
  Hypophysitis: number analyzed (Participants) | 0 | 1 | 0
  Hypophysitis |  | 81.9 [81.9 to 81.9] |

7. Secondary Outcome: Percentage of Participants With a Resolution of IMAEs After Initiating Immune Modulating Medication
Description: Percentage of participants with a resolution of IMAEs after initiating immune modulating medication.
Time Frame: Up to 100 days of the last dose of study drug (Approximately 2 years)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Clear Cell Histology | Non-Clear Cell Histology | Brain Metastasis
Number analyzed (Participants) | 97 | 44 | 1
Percentage of participants
  Pneumonitis: number analyzed (Participants) | 2 | 0 | 0
  Pneumonitis | 100 |  |
  Diarrhea/Colitis: number analyzed (Participants) | 1 | 0 | 0
  Diarrhea/Colitis | 100 |  |
  Hepatitis: number analyzed (Participants) | 5 | 0 | 0
  Hepatitis | 100 |  |
  Adrenal Insufficiency: number analyzed (Participants) | 1 | 0 | 0
  Adrenal Insufficiency | 0 |  |
  Nephritis And Renal Dysfunction: number analyzed (Participants) | 3 | 1 | 0
  Nephritis And Renal Dysfunction | 66.7 | 0 |
  Rash: number analyzed (Participants) | 12 | 2 | 0
  Rash | 83.3 | 50 |
  Hypersensitivity: number analyzed (Participants) | 2 | 0 | 0
  Hypersensitivity | 100 |  |
  Hyperthyroidism: number analyzed (Participants) | 1 | 0 | 0
  Hyperthyroidism | 0 |  |
  Hypophysitis: number analyzed (Participants) | 0 | 1 | 0
  Hypophysitis |  | 0 |

ADVERSE EVENTS:
Time Frame: Adverse events were reported between first dose and 30 days after last dose of study drug: Approximately 4 years and 7 months All Cause Mortality was calculated from first patient first visit to last patient last visit. Approximately 5 years and 4.5 months.
Groups:
- Total: Total Participants
Arm/Group | Clear Cell Histology | Non-Clear Cell Histology | Brain Metastasis | Total
All-Cause Mortality (participants affected / at risk) | 63/97 | 29/44 | 1/1 | 93/142
Serious Adverse Events (participants affected / at risk) | 54/97 | 19/44 | 0/1 | 73/142
Other Adverse Events (participants affected / at risk) | 91/97 | 41/44 | 1/1 | 133/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clear Cell Histology (N=97) | Non-Clear Cell Histology (N=44) | Brain Metastasis (N=1) | Total (N=142)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1 | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Asthenia (General disorders) | 1 | 1 | 0 | 2
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0 | 0 | 1
Norovirus infection (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 1 | 0 | 5
Sepsis (Infections and infestations) | 2 | 2 | 0 | 4
Septic shock (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 | 0 | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 11 | 0 | 29
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Tumour pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 1
Intracranial mass (Nervous system disorders) | 1 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 3 | 2 | 0 | 5
Nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
Peripheral embolism (Vascular disorders) | 0 | 1 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clear Cell Histology (N=97) | Non-Clear Cell Histology (N=44) | Brain Metastasis (N=1) | Total (N=142)
Anaemia (Blood and lymphatic system disorders) | 19 | 5 | 0 | 24
Ear pain (Ear and labyrinth disorders) | 2 | 3 | 0 | 5
Hyperthyroidism (Endocrine disorders) | 8 | 2 | 0 | 10
Hypothyroidism (Endocrine disorders) | 9 | 3 | 0 | 12
Vision blurred (Eye disorders) | 4 | 1 | 1 | 6
Abdominal distension (Gastrointestinal disorders) | 4 | 6 | 0 | 10
Abdominal pain (Gastrointestinal disorders) | 11 | 5 | 0 | 16
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2 | 0 | 8
Constipation (Gastrointestinal disorders) | 25 | 13 | 0 | 38
Diarrhoea (Gastrointestinal disorders) | 18 | 8 | 0 | 26
Dry mouth (Gastrointestinal disorders) | 8 | 2 | 0 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 5 | 0 | 8
Nausea (Gastrointestinal disorders) | 23 | 17 | 0 | 40
Stomatitis (Gastrointestinal disorders) | 5 | 0 | 0 | 5
Vomiting (Gastrointestinal disorders) | 18 | 6 | 0 | 24
Asthenia (General disorders) | 8 | 3 | 0 | 11
Chills (General disorders) | 5 | 5 | 0 | 10
Fatigue (General disorders) | 41 | 16 | 0 | 57
Non-cardiac chest pain (General disorders) | 7 | 0 | 0 | 7
Oedema peripheral (General disorders) | 14 | 5 | 0 | 19
Pain (General disorders) | 6 | 4 | 0 | 10
Pyrexia (General disorders) | 9 | 5 | 1 | 15
Nasopharyngitis (Infections and infestations) | 5 | 1 | 0 | 6
Sinusitis (Infections and infestations) | 5 | 0 | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 13 | 5 | 0 | 18
Urinary tract infection (Infections and infestations) | 13 | 5 | 0 | 18
Alanine aminotransferase increased (Investigations) | 7 | 1 | 0 | 8
Aspartate aminotransferase increased (Investigations) | 8 | 2 | 0 | 10
Blood alkaline phosphatase increased (Investigations) | 5 | 2 | 0 | 7
Blood creatinine increased (Investigations) | 17 | 1 | 0 | 18
Blood thyroid stimulating hormone increased (Investigations) | 4 | 3 | 0 | 7
Weight decreased (Investigations) | 13 | 6 | 0 | 19
Weight increased (Investigations) | 8 | 2 | 0 | 10
Decreased appetite (Metabolism and nutrition disorders) | 25 | 9 | 0 | 34
Dehydration (Metabolism and nutrition disorders) | 8 | 5 | 0 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 3 | 0 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4 | 0 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 3 | 0 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 12 | 0 | 36
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 16 | 0 | 38
Flank pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 0 | 9
Groin pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14 | 4 | 0 | 18
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 1 | 0 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 3 | 0 | 16
Dizziness (Nervous system disorders) | 10 | 4 | 0 | 14
Headache (Nervous system disorders) | 8 | 5 | 1 | 14
Anxiety (Psychiatric disorders) | 8 | 3 | 0 | 11
Confusional state (Psychiatric disorders) | 6 | 0 | 0 | 6
Depression (Psychiatric disorders) | 8 | 1 | 0 | 9
Insomnia (Psychiatric disorders) | 13 | 3 | 1 | 17
Haematuria (Renal and urinary disorders) | 8 | 4 | 0 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 13 | 0 | 38
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 7 | 0 | 23
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 0 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 0 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 2 | 0 | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 11 | 0 | 27
Rash (Skin and subcutaneous tissue disorders) | 14 | 3 | 0 | 17
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 1 | 0 | 6
Rash pruritic (Skin and subcutaneous tissue disorders) | 9 | 1 | 0 | 10
Hypertension (Vascular disorders) | 5 | 2 | 0 | 7
Hypotension (Vascular disorders) | 2 | 3 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/35/NCT02596035/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT02596035/SAP_001.pdf